CLINICAL TRIAL: NCT03892356
Title: Oculomotor Function Testing in Patients Who Suffered Concussions
Brief Title: Oculomotor Function Testing in Acute Concussion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Carmela Tartaglia, Marion and Gerald Soloway Chair in Brain Injury and Concussion Research Associate Professor, University of Toronto, University Health Network, Toronto
Other Study IDs: 18-6196
Record Dates: First submitted 2019-03-21; First posted 2019-03-27 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Concussion, Brain
Keywords: Concussion, Oculomotor function
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Concussion Group: Participants (age group 18-60) who presents to the emergency department in the University Health Network within 7 days of concussion
- Healthy Controls Group: Participants (age group 18-60) with no previous history of concussions who are age, education and sex-matched to the patients' group will be recruited from the community.

SUMMARY:
This is a prospective longitudinal study which aims to compare oculomotor function and visual scanning behaviour (VSB) of participants who suffered concussion with healthy controls with no concussion. This study also aims to investigate the pattern of change in oculomotor function and visual scanning behaviour (VSB) in the participants over a 6-month period.

DETAILED DESCRIPTION:
Primary Objective

* To identify differences in oculomotor function and visual scanning behaviour (VSB) between participant with and without acute concussion
* To investigate patterns of change and recovery in oculomotor function and VSB in participants who suffered a concussion

Secondary Objective

• To investigate the association between the oculomotor function and concussion-related symptoms

This is a prospective longitudinal study which aims to evaluate differences in oculomotor function and visual scanning behaviour (VSB) between participants who suffered acute concussion and healthy controls with no concussion. This study also aims to investigate the pattern of change in oculomotor function and visual scanning behaviour (VSB) in the participants over a 6-month period.

Health information and concussion history: After obtaining informed consents, during the first visit, participants will be asked about their health history such as past medical history, medication history, substance use history, and family history. They will also be asked about their concussion history which includes number of concussions in the past, any comorbidity with the concussions, mechanism of injury, and any change in their levels of consciousness at the time of concussion.

Self-reported outcomes: During each visit, participants will be asked on the presence or absence of concussion-related symptoms and the extent to which these symptoms affect their everyday functioning if present. The symptoms the participants will be questioned using the Rivermead Post-concussive Symptom Questionnaire (RPQ) as a standardized assessment (https://www.commondataelements.ninds.nih.gov/TBI.aspx#tab=Data_Standards) at each visit .

Oculomotor function testing and visual scanning behaviour (VSB): During each visit, oculomotor data will be collected using Visual Attention Scanning Technology (VAST, EL-MAR Inc.). VAST is a technology that was developed to support advanced eye-tracking research application. Over the past 10 years the technology has been used in research studies in the University of Toronto, and University Health Network hospitals. Participants will be seated 65 cm from the monitor, and their binocular gaze positions will be estimated 30 times/sec with an accuracy of 0.5º in visual angle. Following a calibration procedure, the participants will be instructed to look at a series of slides presented on the monitor, and their eye positions will be recorded. The eye positions will be segmented into fixations that are linked to the displayed images. Oculomotor functions testing includes testing self-paced saccadic (SPS) eye movements, fixation, anti-saccadic eye movements. Visual scanning behaviour (VSB) will be assessed using a set of images which require patients to look at the images and match them according to the instruction at the beginning of each test.

Patients will be assessed at baseline (i.e. within 7 days of concussion) and three follow-up (f/u) visits (i.e. 1, 3, and 6 months after concussion).

Healthy controls will be assessed at baseline and one follow-up visit (i.e. 6 months after the baseline).

The entire assessment in each visit takes 30-45 minutes.

ELIGIBILITY:
Concussion Patients:

Inclusion Criteria:

• Participants (age group 18-60) who present to the emergency department in the University Health Network within 7 days of concussion

Exclusion Criteria:

* Age less than 18
* Any other neurological disorder (e.g. seizures)
* Any systemic illness known to affect the brain (e.g. diabetes and lupus)
* History of major psychiatric disorder (e.g. bipolar, schizophrenia)
* History of known developmental disorders (e.g. attention deficit disorder, dyslexia)
* Any lesion detected by MRI prior to the study
* Any previous vision disorder that prevents the participant from performing the self-paced saccade task
* Any brain injury more severe than concussion

Controls:

• Participants (age group 18-60) with no previous history of concussions who are age, education and sex-matched to the patients' group will be recruited from the community.

Healthy Controls:

Inclusion Criteria:

• Participants (age group 18-60) with no previous history of concussions who are age, education and sex-matched to the patients' group will be recruited from the community.

Exclusion Criteria:

• All exclusion criteria mentioned above for patients plus any history of concussions

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: 100 participants who suffered concussions and present to the emergency department in the University Health Network within 7 days of concussion will be compared with 20 healthy volunteers who have no history of concussions.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
self-paced saccade | 2 years
  Number of self paced saccadic eye movements in 60 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Canadian Concussion Centre, Toronto Western Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No